CLINICAL TRIAL: NCT07223671
Title: Phase 1, 2-Cohort, Open-label, Fixed-sequence, Drug-drug Interaction Study to Evaluate the Effect of Repotrectinib on the Pharmacokinetics of Transporter and CYP P450 Probe Substrates in Healthy Adult Participants
Brief Title: Study to Evaluate the Effect of Repotrectinib on the Drug Levels of Transporter and CYP P450 Probe Substrates in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1088
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Drug-Drug Interactions; Pharmacokinetics; Transporter Probe Substrates; CYP P450 Probe Substrates
MeSH Terms: interventions — repotrectinib; Metformin; Digoxin; Rosuvastatin Calcium; Bupropion; Flurbiprofen; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: Repotrectinib; Drug: Metformin; Drug: Digoxin; Drug: Rosuvastatin
- Cohort 2 (Experimental)
  Interventions: Drug: Repotrectinib; Drug: Bupropion; Drug: Flurbiprofen; Drug: Omeprazole

INTERVENTIONS:
Drug: Repotrectinib — Specified dose on specified days
Drug: Metformin — Specified dose on specified days
  Arms: Cohort 1
Drug: Digoxin — Specified dose on specified days
  Arms: Cohort 1
Drug: Rosuvastatin — Specified dose on specified days
  Arms: Cohort 1
Drug: Bupropion — Specified dose on specified days
  Arms: Cohort 2
Drug: Flurbiprofen — Specified dose on specified days
  Arms: Cohort 2
Drug: Omeprazole — Specified dose on specified days
  Arms: Cohort 2

SUMMARY:
The purpose of the study if to evaluate the effect of Repotrectinib on the drug levels of transporter and CYP P450 probe substrates in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria

* Participants must have a body mass index (BMI) of 18.0 to 32.0 kg/m2 and should be between the ages of 18-60 years inclusive.
* Healthy female (as assigned at birth) participants who are individuals not of childbearing potential (INOCBP) and healthy males with no clinically significant deviation from normal for the following: medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory assessment results as determined by the investigator.

Exclusion Criteria

* Participants must not have a significant history of clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, psychiatric, neoplastic, or genitourinary abnormalities/diseases as determined by the investigator or designee.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration of AUC (0-T) of Probe Substrate With Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains metformin, digoxin, and rosuvastatin.
Cohort 1: AUC (0-T) of Probe Substrate Without Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains metformin, digoxin, and rosuvastatin.
Cohort 1: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of Probe Substrate With Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains metformin, digoxin, and rosuvastatin.
Cohort 1: AUC(INF) of Probe Substrate Without Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains metformin, digoxin, and rosuvastatin.
Cohort 1: Maximum Observed Plasma Concentration (Cmax) of Probe Substrate With Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains metformin, digoxin, and rosuvastatin
Cohort 1: Cmax of Probe Substrate Without Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains metformin, digoxin, and rosuvastatin
Cohort 1: Area Under the Plasma Concentration-time Curve From Time Zero to 48 Hours Post Dose (AUC (0-48)) of Metformin With Repotrectinib | Up to approximately Day 17 post dose
Cohort 1: AUC (0-48) of Metformin Without Repotrectinib | Up to approximately Day 17 post dose
Cohort 1: Renal Clearance (CLR) of Metformin in Urine | Up to approximately Day 16 post dose
Cohort 2: AUC (0-T) of Probe Substrate With Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains bupropion, hydroxybupropion, flurbiprofen, 4'-hydroxyflurbiprofen, omeprazole, 5'- hydroxyomeprazole)
Cohort 2: AUC (0-T) of Probe Substrate Without Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains bupropion, hydroxybupropion, flurbiprofen, 4'-hydroxyflurbiprofen, omeprazole, 5'- hydroxyomeprazole)
Cohort 2: AUC (INF) of Probe Substrate With Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains bupropion, hydroxybupropion, flurbiprofen, 4'-hydroxyflurbiprofen, omeprazole, 5'- hydroxyomeprazole)
Cohort 2: AUC (INF) of Probe Substrate Without Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains bupropion, hydroxybupropion, flurbiprofen, 4'-hydroxyflurbiprofen, omeprazole, 5'- hydroxyomeprazole)
Cohort 2: Cmax of Probe Substrate With Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains bupropion, hydroxybupropion, flurbiprofen, 4'-hydroxyflurbiprofen, omeprazole, 5'- hydroxyomeprazole)
Cohort 2: Cmax of Probe Substrate Without Repotrectinib | Up to approximately Day 17 post dose
  Probe substrate contains bupropion, hydroxybupropion, flurbiprofen, 4'-hydroxyflurbiprofen, omeprazole, 5'- hydroxyomeprazole)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately Day 45 post dose
Number of Participants with Serious Adverse Events (SAEs) | Up to approximately Day 45 post dose
Number of Participants With Clinically Significant Physical Examination Findings | Up to approximately Day 17 post dose
Number of Participants With Clinically Significant Vital Sign Measurements | Up to approximately Day 17 post dose
Number of Participants With Clinically Significant 12-lead Electrocardiogram (12-lead ECG) Findings | Up to approximately Day 17 post dose
Number of Participants With Clinically Significant Safety Laboratory Test Results | Up to approximately Day 17 post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Fortrea Clinical Research Unit - Daytona Beach, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Bristol Myers Squibb (BMS) will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding BMS's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07223671.html